CLINICAL TRIAL: NCT02032043
Title: Optimization of Mass Drug Administration With Existing Drug Regimens for Lymphatic Filariasis and Onchocerciasis for Ivory Coast
Brief Title: Optimization of Mass Drug Administration With Existing Drug Regimens for Lymphatic Filariasis and Onchocerciasis for Ivory Coast (DOLF-Ivory Coast)
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Gary Weil, MD, Professor of Medicine/Microbiology, Washington University School of Medicine
Other Study IDs: 201306100
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Lymphatic Filariasis; Onchocerciasis; Soil Transmitted Helminth (STH) Infections
Keywords: Filariasis; Onchocerciasis; Albendazole; Ivermectin; STH Soil Transmitted Helminth infections; MDA Mass Drug Administration
MeSH Terms: conditions — Elephantiasis, Filarial; Onchocerciasis; Infections; Filariasis | interventions — Albendazole; Ivermectin

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Study procedures include collection of finger prick blood that will be tested for microfilaremia and for serology testing (antigenemia and antibody testing). Investigators will also collect skin snips (small superficial skin biopsies) to detect Onchocerca microfilariae, and stool samples to detect parasitic worm eggs indicative of STH infections.
  All assays will be performed in Ivory Coast(filarial serology tests, MF smears, stool examinations).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Annual MDA treated Group: This group will receive annual mass drug administration (Albendazole 400 mg plus Ivermectin) provided by the Ivorian Ministry of Health.
  Interventions: Drug: Annual versus Semiannual Albendazole plus Ivermectin MDA
- Semiannual Mass Drug Administration: This group will receive semi-annual mass drug administration (Albendazole 400 mg plus Ivermectin) provided by the Ivorian Ministry of Health.
  Interventions: Drug: Annual versus Semiannual Albendazole plus Ivermectin MDA

INTERVENTIONS:
Drug: Annual versus Semiannual Albendazole plus Ivermectin MDA — Annual or semiannual Albendazole plus Ivermectin, administered by the Ivorian Ministry of Health.
  Other Names: Albenza (Albendazole); Mectizan (Ivermectin)

SUMMARY:
Approximately 4,000 people will participate per year. The study population will include females and males over 5 years of age who live in filariasis and onchocerciasis endemic areas. Subject selection will not be based on health status.

Two sites will be studied, and each study will last for 4 years. Participants will be studied only once in cross-sectional surveys. Some subjects may be included in more than one annual population survey, but this is not a longitudinal study.

Investigators will compare annual and semiannual mass drug administration (MDA) for lymphatic filariasis and onchocerciasis, and investigators will compare the impact of these MDA schedules on soil transmitted helminth infections. MDA will be administered by others (Ivorian Ministry of Health).

The investigators will test the hypothesis that semiannual mass drug administration (MDA) is superior to annual MDA for elimination of lymphatic filariasis, onchocerciasis and for control of soil transmitted helminth (STH) infections.

1. Compare the relative impact and cost effectiveness of annual vs. twice yearly mass drug administration (MDA) for elimination of lymphatic filariasis (LF) in these populations.
2. Compare the relative impact and cost effectiveness of annual vs. twice yearly mass drug administration (MDA) for elimination of onchocerciasis in these populations.
3. Study the impact of annual vs. semiannual MDA on soil transmitted helminth (STH) infection in these populations.

DETAILED DESCRIPTION:
Lymphatic filariasis (LF) is a deforming and disabling infectious disease that causes elephantiasis and genital deformity (especially hydroceles). The infection affects some 120 million people in 81 countries in tropical and subtropical regions with well over 1 billion people at risk of acquiring the disease [1]. LF is caused by Wuchereria bancrofti and Brugia spp. (B. malayi and B.timori), nematode parasites that are transmitted by mosquitoes. This study is based on the assumption that currently used MDA regimens and schedules are not optimal for achieving elimination of LF. These regimens (either annual Albendazole (Alb) 400 mg plus diethylcarbamazine 6 mg/kg or Alb 400 mg plus Ivermectin (Iver) 200 µg/kg for LF) were introduced more than 10 years ago.

Onchocerciasis ("Oncho") is similar in some ways to LF in that it is a vector-borne nematode parasitic disease that causes severe disability. In contrast to LF, this disease causes blindness and severe skin disease rather than elephantiasis, and it is spread by black flies instead of mosquitoes. O. volvulus adult worms live in subcutaneous nodules while the adult worms of the LF parasites live in lymphatic vessels. O. volvulus adult worms are larger and less sensitive to available drug treatments than those of the species that cause LF and have a longer lifespan (approximately 14 years rather than the estimated 7 years for LF parasites). More effective drugs or dosing schedules for MDA against Oncho could shorten the number of years needed to interrupt Oncho transmission in areas that previously had high disease rates.

Drugs used for LF MDA are also active against soil transmitted helminth infections (STH, e.g., Ascaris, Hookworm, and Trichuris). De-worming campaigns using anthelmintics usually target special groups of the population, such as schoolchildren, and have limited impact on transmission. Treatment of the total population and semiannual treatments may reduce re-infection considerably and will most likely lead to reduced infection densities and infection prevalence rates. Suppression of STH is an important ancillary benefit of MDA programs for filarial infections. Increasingly control programs for filariasis and STH are being integrated with programs for other parasitic diseases such as schistosomiasis. For this reason, participants will also be tested for schistosomiasis.

Purpose: The study aims to compare the effectiveness once yearly (1X) versus twice yearly (2X) mass drug administration (MDA) for the elimination of lymphatic filariasis, onchocerciasis and for control of soil-transmitted helminth infections (intestinal parasites) in large populations. Mass drug administration will be provided by the Ivory Coast Ministry of Health. This project will assess the impact of the government's public health program.

Procedures: Study procedures include collection of finger prick blood that will be tested for microfilariae by microscopy and for serology testing (antigenemia and antibody testing). Skin snips will be collected and examined by microscopy for the presence of Onchocerca microfilariae. Stool samples will be collected for detection of parasitic worm eggs by microscopy. All assays will be performed in Ivory Coast(filarial serology tests, microfilaria testing, stool examinations).

Washington University researchers developed the protocol, will provide training and guidance to Ivorian researchers, and work with them to analyze the data. Ivorian researchers will consent the participants, obtain blood, skin and stool specimens, perform laboratory tests on the specimens, and enter data on participants and lab results.

ELIGIBILITY:
Inclusion Criteria:

* Study areas should be endemic for filariasis and onchocerciasis.
* Study population have limited or no prior experience with MDA. Males and Females greater than or equal to 5 years of age.

Exclusion Criteria:

* Children less than 5 years of age.
* Children who weigh less than 15 kg (33 lb)

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study populations are people who live in areas of Ivory Coast that are co-endemic for lymphatic filariasis and onchocerciasis.
Sampling Method: Probability Sample
Enrollment: 14457 (Actual)
Dates: Start 2014-02; Primary Completion 2017-12-04 (Actual); Study Completion 2017-12-04 (Actual)

PRIMARY OUTCOMES:
Microfilaria prevalence based on results of microscopic examination of blood smears and skin snips. | 4 years
  From annual population based surveys, the prevalence of microfilaremia (filarial parasites in the blood or skin snips) will be assessed by microscopic examination of slides with thick blood smears and skin snips. Test results for individuals are either positive or negative. The unit for prevalence studies is the percentage (%) of individuals with positive tests.

SECONDARY OUTCOMES:
Prevalence of filarial antigenemia in blood and intensity of filarial and intestinal worm infections based on results of microscopy. | 4 years
  Secondary outcomes for the study include prevalence of filarial antigenemia (detected with the Alere Filariasis Strip test) and prevalence of worm eggs in stool detected by the Kato-Katz test. Both of these outcomes are qualitative with no units of measure (positive or negative). Other secondary outcome measures will be intensity of infection by counting microfilaria (Mf) in blood (Mf per ml of blood) and counting Mf in skin (Mf per milligram) and by counting worm eggs (eggs per gram of stool, assessed separately for each parasite species). All of these quantitative assessments are based on counting parasites by microscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Gary J Weil, MD, Principal Investigator — Washington University School of Medicine; Peter U Fischer, PhD, Principal Investigator — Washington University School of Medicine; Aboulaye Miete, MD, Study Director — Ivory Coast Ministry of Health, National Program Against Filariasis, Schistosomiasis and Geohelminths
Locations (1):
- Ivory Coast National Program Against Schistosomiasis, Geohelminths and Filariasis, Abidjan, Lagune-Cocody, Côte d’Ivoire

REFERENCES:
- [Derived] Loukouri A, Meite A, Koudou BG, Goss CW, Lew D, Weil GJ, N'Goran EK, Fischer PU. Impact of annual and semi-annual mass drug administration for Lymphatic Filariasis and Onchocerciasis on Hookworm Infection in Cote d'Ivoire. PLoS Negl Trop Dis. 2020 Sep 25;14(9):e0008642. doi: 10.1371/journal.pntd.0008642. eCollection 2020 Sep. PMID 32976514
- See also: Death to Onchocerciasis and Lymphatic Filariasis (DOLF) Project — http://www.dolf.wustl.edu/